CLINICAL TRIAL: NCT00648258
Title: A Double-Blind, Double Dummy, Randomized Comparison Study Of The Efficacy And Safety Of Valdecoxib 10mg QD And Naproxen 500mg BID In Treating The Signs And Symptoms Of Osteoarthritis Of The Knee Or Hip In Taiwan
Brief Title: A Double-Blind, Double Dummy, Randomized Comparison Study Of The Efficacy And Safety Of Valdecoxib 10mg Once Daily And Naproxen 500mg Twice Daily In Treating The Signs And Symptoms Of Osteoarthritis Of The Knee Or Hip In Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VALA-0513-141; A3471101
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, knee; osteoarthritis, hip
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — valdecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: naproxen

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 10 mg tablet by mouth once daily for 6 weeks
  Arms: Arm 1
Drug: naproxen — naproxen 500 mg capsule by mouth twice daily for 6 weeks
  Arms: Arm 2

SUMMARY:
To evaluate the efficacy, safety, and tolerability of valdecoxib by comparing valdecoxib 10 mg daily (QD) with naproxen 500 mg twice daily (BID) in treating the signs and symptoms of osteoarthritis (OA) of the knee or hip. The study was designed to collect comparative information for the local population (Taiwan).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of hip OA, which was having hip pain and meeting criteria for at least 2 of the following: a. Westergren erythrocyte sedimentation rate of < 20 mm/hr; b. radiographic femoral or acetabular osteophytes or c. radiographic joint space narrowing
* Knee OA diagnosis required diagnosing (by modified American College of Rheumatology criteria) OA of the knee with pain plus at least one of the following: a. Age> 50 years old, b. Stiffness < 30 minutes, c. crepitus on active motion and radiographic evidence of OA of the knee, defined as presence of osteophytes or joint space narrowing
* Symptomatic OA of the knee or hip was determined at the Baseline Visit, if the Patient's Assessment of Arthritis Pain was at least 40 mm VAS, Patient's and the Physician's Global Assessment of Arthritis was "poor" or "very poor"

Exclusion Criteria:

* Use of NSAIDs or analgesics within 2 days (within 4 days for subjects taking oxaprozin, piroxicam or full dose aspirin) before baseline arthritis assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2003-07; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Patient's Assessment of Arthritis Pain (Osteoarthritis-Pain VAS) | Week 6

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC OA) Composite Index | Week 2 and Week 6
WOMAC OA physical function | Week 2 and Week 6
WOMAC OA pain index | Week 2 and Week 6
WOMAC OA stiffness index | Week 2 and Week 6
Patient's Assessment of Arthritis Pain (Osteoarthritis-Pain VAS) | Week 2
Patient's Global Assessment of Arthritis | Week 2 and Week 6
Physician's Global Assessment of Arthritis | Week 2 and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Taiwan (4):
  - Pfizer Investigational Site, Kweishan, Taoyuan
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taichung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALA-0513-141&StudyName=A%20Double-Blind%2C%20Double%20Dummy%2C%20Randomized%20Comparison%20Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20Valdecoxib%2010mg%20QD%20And%20Naproxen%20500mg%20BID%20In%20Treating%20The%20Signs%20And%20Symptoms%20Of%20Osteoarthritis%20Of%20The%20Knee%20Or%20Hip%20In%20Taiwan